CLINICAL TRIAL: NCT03524586
Title: Comparison of the Endotracheal Tube Cuff Pressure of a Taper-guard Cuffed Tube Between Ipsilateral and Contralateral Rotation of Head During Tympanoplasty; Prospective Study.
Brief Title: Comparison of the Cuff Pressure of a Taper-guard Cuffed Tube Between Ipsilateral and Contralateral Rotation of Head
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Saeyoung Kim, MD, PhD, Associate professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2017-12-001-002
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Anesthesia, Endotracheal; Airway Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ipsilateral rotation of head (Experimental): Head was laterally rotated to the same side against fixed tube
  Interventions: Procedure: Ipsilateral rotation of head
- Contralateral rotation of head (Active Comparator): Head was laterally rotated to the opposite side against fixed tube
  Interventions: Procedure: Contralateral rotation of head

INTERVENTIONS:
Procedure: Ipsilateral rotation of head — Ipsilateral rotation of head against fixed tube
  Arms: Ipsilateral rotation of head
Procedure: Contralateral rotation of head — Contralateral rotation of head against fixed tube
  Arms: Contralateral rotation of head

SUMMARY:
This study evaluates the endotracheal tube cuff pressure of a taper-guard cuffed tube during tympanoplasty with ipsilateral rotation of head, compared to the contralateral rotation of head.

The investigators will performed the ipsilateral rotation of head against the fixed tube in half of participants or the contralateral rotation of head in the other half.

DETAILED DESCRIPTION:
The inflation of the endotracheal tube cuff is very useful to prevent aspiration of contaminated substances into lung past endotracheal tube and leakage of gas during positive pressure ventilation. However, excessive inflation of endotracheal tube cuff frequently causes tracheal mucosal damage, which can increase the incidence of sore throat, hoarseness, and coughing after surgery.

Taper-guard cuffed tube was newly developed. Taper-guard endotracheal tube is more effective in providing a sealing effect than a cylindrical endotracheal tube in an in vitro study. However, recently, it was reported that the cuff pressure of a Taper-guard endotracheal tube significantly increased after a positional change from the supine to the lateral flank position, compared to that of a cylindrical endotracheal tube. However, during tympanoplasty, the investigators need to rotate head for proper position.

In this study, therefore, the investigators investigate the difference of the endotracheal tube cuff pressure of a taper-guard cuffed tube between ipsilateral and contralateral rotation of head against the fixed tube during tympanoplasty.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status classification I-III for a tympanoplasty under general anesthesia

Exclusion Criteria:

* history of difficult intubation, limited neck movement, respiratory diseases, and body mass index >35kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
The endotracheal tube cuff pressure | During procedure
  The endotracheal tube cuff pressure was checked using a manometer

SECONDARY OUTCOMES:
The distance from the endotracheal tube tip to the carina | During procedure
  The distance from the endotracheal tube tip to the carina was recorded again using a fiberoptic bronchoscope.

CONTACTS AND LOCATIONS:
Overall Officials: Saeyoung Kim, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook national university hospital, Daegu, South Korea